CLINICAL TRIAL: NCT02391155
Title: Follicular Flushing Outcomes in Singles Versus Double Lumen Oocyte Retrieval Needles in Poor Responding Patients:a Randomized Controlled Trial
Brief Title: Follicular Flushing Outcomes in Singles Versus Double Lumen Oocyte Retrieval Needles in Poor Responding Patients
Acronym: needles(opu)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Bulent Haydardedeoglu, Assoc. Prof. M.D. Bulent Haydardedeoglu, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KA13/161
Record Dates: First submitted 2015-02-11; First posted 2015-03-18 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2015-03

CONDITIONS: Infertility
Keywords: follicular flushing; IVF; poor responders; oocyte retrival
MeSH Terms: conditions — Infertility | interventions — Oocyte Retrieval

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- single lumen (Active Comparator): Single lumen needle in oocyte retrieval
  Interventions: Procedure: single lumen needle in oocyte retrieval; Procedure: double lumen needle in oocyte retrieval
- double lumen (Active Comparator): Double lumen needle with follicle flushing during oocyte retrieval
  Interventions: Procedure: single lumen needle in oocyte retrieval; Procedure: double lumen needle in oocyte retrieval

INTERVENTIONS:
Procedure: single lumen needle in oocyte retrieval — single lumen needle use during oocyte retrieval
Procedure: double lumen needle in oocyte retrieval — after aspiration of follicles, 3 times flushing will be performed in double lumen needle.

SUMMARY:
In this study, the investigators aimed to evaluate to the efficacy of the needle type used in follicular flushing in oocyte retrieval in the poorest responders undergoing IVF.

DETAILED DESCRIPTION:
This study will include:

1. women with less than four follicles on the day of hCG administration
2. women between 20-45 age old
3. The value of progesterone on the day of hCG administration will be under 1.5ng/ml

ELIGIBILITY:
Inclusion Criteria:

1. women between 20-45 years old
2. the number of follicles less than 5 on the day of HCG administration
3. the value of progesteron on the day of hCG administration must be under 1.5ng/ml

Exclusion Criteria:

1. women under 20 years and older than 45 year
2. on the day of hCG administration if the follicle number is more than 5
3. if.the value of progesteron on the day of hCG administration is higher than 1.5ng/ml

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
number of metaphase 2 oocyte | Six months

SECONDARY OUTCOMES:
clinical pregnancy rate | eigth months

CONTACTS AND LOCATIONS:
Locations (1):
- Bulent Haydardedeoglu, Adana, Turkey (Türkiye)